CLINICAL TRIAL: NCT02248857
Title: Promoting the Universal Medication Schedule Via Mobile and EHR Technologies: A Physician-randomized Control Trial
Brief Title: Promoting the Universal Medication Schedule Via Mobile and EHR Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00097744
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes
Keywords: UMS; medication schedule; diabetes; drug labeling
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Employ the current standard of care. No intervention.
- UMS strategy (Experimental): Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions.
  1. Prescription instructions will be adapted to UMS to establish four standard time intervals for prescribing and dispensing of medicine. UMS instructions also use simplified text and numeric characters instead of words to detail dose.
  2. Single-page, plain language medication information sheets with content from a patient's perspective and following health literacy best practices.
  3. A list of their current medications each corresponding to a set of instructions and a checkbox for morning, noon, evening, and bedtime medicine to help patients visually depict when to take their medicines.
  Interventions: Other: UMS Strategy
- UMS strategy + SMS texting reminders (Experimental): In addition to the components from the UMS strategy arm, patients will receive daily text reminders for 7 days, with the option of extending reminders, following a study medication prescription.
  Interventions: Other: UMS Strategy; Other: SMS Texting Reminders

INTERVENTIONS:
Other: UMS Strategy — Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions.
  Arms: UMS strategy; UMS strategy + SMS texting reminders
Other: SMS Texting Reminders — In addition to the components from the UMS strategy arm, patients will receive daily text reminders for 7 days, with the option of extending reminders, following a study medication prescription.
  Arms: UMS strategy + SMS texting reminders

SUMMARY:
The purpose of this study test the effectiveness of the Universal Medication Schedule (UMS), which was designed as a strategy to standardize and simplify medication instructions to support safe and effective prescription drug use among diabetic.

DETAILED DESCRIPTION:
Research has shown the UMS (1) improves patients' understanding of how much to take of a medicine and when, and (2) reduces the number of times per day patients would take a multi-drug regimen. In this study, UMS tools will be exported into a second electronic health record platform to demonstrate ease of dissemination. Also, as patients may require assistance outside of clinic visits to adapt their prescription regimen to the UMS, this study will test the potential benefit of daily short message service (SMS) text reminders via cell phone.

We will conduct a three-arm, provider-randomized controlled trial among English and Spanish-speaking adults taking three or more prescription drugs to evaluate the effectiveness of the UMS strategy, with and without SMS text reminders, to improve patient understanding, consolidation, and adherence compared to usual care.We will conduct a three-arm, provider-randomized trial at two community health centers in Chicago, IL to evaluate the UMS and UMS+SMS text reminder strategies compared to usual care. English and Spanish-speaking patients who are prescribed three or more medications will be recruited and assessed by phone at baseline, three months, and six months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type II diabetes
* age 30 or older
* taking 3 or more prescription medications for chronic conditions
* English or Spanish speaking

Exclusion Criteria:

* self-reported severe, uncorrectable vision
* hearing impairment
* cognitive impairment
* not responsible for administering his/her own medications
* not able to receive text messages on their cell phone

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolf, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Started | 157 | 168 | 127
Completed | 157 | 168 | 127
Not Completed | 0 | 0 | 0
Period: 3 Month
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Started | 157 | 168 | 127
Completed | 111 | 134 | 96
Not Completed | 46 | 34 | 31
Not completed — Withdrawal by Subject | 9 | 3 | 4
Not completed — Unable to reach for 3 month | 35 | 29 | 26
Not completed — Partially completed, unable to finish | 2 | 2 | 1
Period: 6 Month
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Started (Participants were still eligible for the 6 month if they did not complete the 3 month.) | 148 (157 baseline - 9 who withdrew = 148) | 165 (168 baseline - 3 who withdrew = 165) | 123 (127 baseline - 4 who withdrew = 123)
Completed | 120 | 136 | 106
Not Completed | 28 | 29 | 17
Not completed — Lost to Follow-up | 27 | 26 | 15
Not completed — Partially completed, unable to finish | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders | Total
Number analyzed (Participants) | 157 | 168 | 127 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 131 | 142 | 95 | 368
  >=65 years | 26 | 26 | 32 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.4) | 56.4 (9.3) | 57.5 (9.9) | 56.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 108 | 87 | 295
  Male | 57 | 60 | 40 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 113 | 127 | 91 | 331
  Not Hispanic or Latino | 43 | 41 | 36 | 120
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 3 | 6 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 27 | 23 | 82
  White | 112 | 130 | 96 | 338
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 8 | 4 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 157 | 168 | 127 | 452

OUTCOME MEASURES:

1. Primary Outcome: Prescription Understanding
Description: Predictive probabilities of prescription understanding will be calculated based on patients' ability to correctly dose their prescription medications using unadjusted Generalized Estimating Equation models, specifying the binomial family and logit link, with medication as the unit of analysis. Correct dosing per medication will be scored as yes or no, reflecting having demonstrated all of the following: proper dose (# of pills), spacing (hours between doses), frequency (# of times per day), and total pills per day. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after baseline
Population: All participants who completed the 6 month assessment and had complete data for the outcome for at least 1 medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability
Units Other Than Participants: Medications
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 120 | 134 | 104
Number analyzed (Medications) | 559 | 611 | 455
Probability | 0.81 [0.77 to 0.84] | 0.82 [0.79 to 0.85] | 0.78 [0.74 to 0.82]

2. Secondary Outcome: Medication Knowledge
Description: Predictive probabilities of medication knowledge will be calculated based on patients' ability to identify each medication's purpose and side effects, risks, warnings, and benefits using unadjusted Generalized Estimating Equation models, specifying the binomial family and logit link, with medication as the unit of analysis. Patients will be asked through a structured questionnaire about each of the above via structured, open-ended items. Each medication will be scored as correct/incorrect if the participant knew the purpose and could name at least 1 side effect, risk, or warning of the medication. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after baseline
Population: All participants who completed the 6 month assessment and had complete outcome data for at least 1 medication
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of medication knowledge
Units Other Than Participants: Medications
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 120 | 137 | 104
Number analyzed (Medications) | 611 | 654 | 488
Probability of medication knowledge | 0.21 [0.18 to 0.25] | 0.28 [0.25 to 0.32] | 0.26 [0.22 to 0.30]

3. Secondary Outcome: Medication Adherence: Pill Count
Description: Predictive probabilities of medication adherence will be calculated based on telephone pill counts using unadjusted Generalized Estimating Equation models, specifying the binomial family and logit link, with medication as the unit of analysis. Pills taken/pills prescribed will be calculated for each medication and scored as adherent for that medication if that score is between 80% and 120%. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after baseline
Population: All participants who completed the 6 month assessment and had complete outcome data for at least 1 medication
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence
Units Other Than Participants: Medications
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 109 | 128 | 98
Number analyzed (Medications) | 296 | 366 | 277
Probability of adherence | 0.41 [0.35 to 0.47] | 0.31 [0.27 to 0.36] | 0.34 [0.29 to 0.40]

4. Secondary Outcome: Medication Adherence: PMAQ
Description: Predictive probabilities of medication adherence will be calculated based on a 4-item validated Patient Medication Adherence Questionnaire (PMAQ) using unadjusted Generalized Estimating Equation models, specifying the binomial family and logit link, with medication as the unit of analysis. The PMAQ assesses adherence behaviors by asking patients to self-report missed/wrong doses in past 4 days, scoring each medication as adherent for that medication if no missed doses were reported. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after baseline
Population: All participants who completed the 6 month assessment and had complete outcome data for at least 1 medication
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence
Units Other Than Participants: Medications
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 120 | 137 | 104
Number analyzed (Medications) | 609 | 654 | 487
Probability of adherence | 0.71 [0.68 to 0.75] | 0.72 [0.69 to 0.76] | 0.77 [0.73 to 0.81]

5. Secondary Outcome: Medication Adherence: Pharmacy Records
Description: Predictive probabilities of primary medication adherence will be calculated based on the proportion of days covered (PDC) with medication obtained from pharmacy records using unadjusted Generalized Estimating Equation models, specifying the binomial family and logit link, with medication as the unit of analysis. PDC is calculated by summing the number of days' supply obtained by a patient during a given time period and dividing by the number of days for which the patient was prescribed the medication. Each medication is scored as adherent if the patient was covered for that medication more than 80% of the time. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after baseline
Population: Participants who filled medications at Walgreens during the study period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence
Units Other Than Participants: Medications
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 33 | 45 | 33
Number analyzed (Medications) | 168 | 217 | 177
Probability of adherence | 0.49 [0.41 to 0.57] | 0.59 [0.52 to 0.65] | 0.55 [0.48 to 0.63]

6. Other Pre Specified Outcome: Changes in Blood Pressure
Description: An exploratory analysis will be conducted to investigate the impact of receiving the UMS in either intervention arm on biologic outcomes for these prevalent conditions. Systolic blood pressure will be obtained from patients' electronic health records. Differences will be measured between the last clinical measurement prior to baseline assessment and the last measured value during the study period (closest to 6 month assessment).
Time Frame: 6 months before baseline to 1 year after baseline
Population: All participants with both a baseline and 6 month systolic blood pressure measurement
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 94 | 115 | 91
mmHG | -1.4 (14.1) | 0.5 (14.0) | 0.1 (15.5)

7. Other Pre Specified Outcome: Changes in Hemoglobin A1c (hbA1c)
Description: An exploratory analysis will be conducted to investigate the impact of receiving the UMS in either intervention arm on biologic outcomes for these prevalent conditions. Hemoglobin A1c (hbA1c) will be obtained from patients' electronic health records. Differences will be measured between the last clinical measurement prior to baseline assessment and the last measured value during the study period (closest to 6 month assessment).
Time Frame: 6 months before baseline to 1 year after baseline
Population: All participants with both a baseline and 6 month hbA1c measurement
Measure: Mean (Standard Deviation); unit: percent of glycated hemoglobin
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 114 | 136 | 105
percent of glycated hemoglobin | -0.2 (1.3) | -0.1 (1.5) | -0.2 (1.4)

8. Other Pre Specified Outcome: Changes in Low-density Lipoprotein Cholesterol (LDL)
Description: An exploratory analysis will be conducted to investigate the impact of receiving the UMS in either intervention arm on biologic outcomes for these prevalent conditions. Low-density lipoprotein cholesterol (LDL) will be obtained from patients' electronic health records. Differences will be measured between the last clinical measurement prior to baseline assessment and the last measured value during the study period (closest to 6 month assessment).
Time Frame: 6 months before baseline to 1 year after baseline
Population: All participants with both a baseline and 6 month LDL measurement
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Number analyzed (Participants) | 19 | 29 | 9
mg/dL | -10.1 (26.7) | -17.1 (66.5) | -23.4 (38.7)

ADVERSE EVENTS:
Arm/Group | Usual Care | UMS Strategy | UMS Strategy + SMS Texting Reminders
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/168 | 0/127
Other Adverse Events (participants affected / at risk) | 0/157 | 0/168 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No